CLINICAL TRIAL: NCT01663662
Title: The Use of Tolvaptan to Prevent Renal Dysfunction in High Risk Patients With Acute Decompensated Heart Failure-Pilot Study
Brief Title: The Use of Tolvaptan to Prevent Renal Dysfunction in High Risk Patients With Heart Failure-Pilot Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of eligible patients
Sponsor: University of Michigan (Other)
Collaborators: Otsuka Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Barry E. Bleske, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-PAF06621
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan Arm (Active Comparator): Tolvaptan 30 mg qd x 3 days and Low Dose Loop Continuous Infusion - Initial Dosing:
  Furosemide - 10 mg/hr Bumentanide - 0.25 mg/hr Torsemide - 5 mg/hr
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Placebo x 3 days and standard of care continuous infusion diuretic
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tolvaptan
  Arms: Tolvaptan Arm
Drug: placebo
  Arms: Placebo

SUMMARY:
It is well known that the use of loop diuretics in acute setting may decrease glomerular filtration rate (GFR) and increase serum creatinine leading to renal dysfunction. Loop diuretic induced elevation in serum creatinine can lead to increase in length of hospital stay and possibly morbidity. Previous studies have suggested that tolvaptan unlike aggressive loop diuretic therapy may not activate neurohormonal system nor decrease renal blood flow. These properties may make tolvaptan a useful addition to diuretic therapy to prevent renal dysfunction in high-risk patients. Therefore the primary objective of this study is to determine if the use of tolvaptan in combination with diuretic therapy may prevent development of renal dysfunction in high risk patients with heart failure.

Hypothesis: Administration of tolvaptan in combination with continuous loop diuretic therapy in acutely decompensated heart failure patients at high risk for developing diuretic induced renal dysfunction will have a lower proportion of patients increasing their serum creatinine > 0.3 mg/dL within a 96 hour time frame as compared to patients just receiving standard of care continuous infusion diuretic.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Prior clinical diagnosis of systolic heart failure (EF < 40% within the past 18 months) with daily home use of oral loop diuretic for at least one month.
* Daily oral dose of furosemide ≥ 40 mg and ≤ 240 mg (or equivalent)
* Identified within 24 hours of hospital admission
* Heart failure defined by at least 1 symptom (dyspnea, orthopnea, or edema) AND 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography)
* Anticipated need for IV loop diuretics for at least 48 hours
* Likely requires daily net urine output in the range of 1-3 L/day for over a 72-96 hour time period.
* Albumin level < 3.5 g/dL
* Willingness to provide informed consent

Exclusion Criteria:

* Received or planned IV vasoactive treatment (inotropes, vasodilators) or ultra-filtration therapy for heart failure
* BNP < 250 ng/ml or NT-proBNP < 1000 mg/ml (if drawn for clinical purposes)
* Systolic BP < 90 mmHg
* Serum creatinine > 3.0 mg/dl at baseline or renal replacement therapy or creatinine clearances < 10 mL/min
* Serum sodium > 145 mEq/L
* Acute coronary syndrome within 4 weeks
* Anticipated need for coronary angiography or other procedures requiring IV contrast.
* Patients receiving any of the following drugs: clarithromycin, ketoconazole, itraconazole,ritonavir, indinavir, nelfinavir, saquinavir, nefazodone, telithromycin, erythromycin, fluconazole, aprepitant, diltiazem, verapamil, cyclosporine, and grapefruit juice.
* Pregnant or nursing patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Renal dysfunction | 96 hours
  Increase in serum creatinine > 0.3 mg/dL within a 96 hours from enrollment

SECONDARY OUTCOMES:
Weight | 24, 78, 72, 96
  Change in weight over 24, 48, 72, and 96 hours
Urine output | 24, 48, 72, 96
  Net urine output over 24, 48, 72, and 96 hours
Hospitalization length of stay | 10

OTHER OUTCOMES:
Treatment Failure | 72hr
  Need to increase diuretic dose in tolvaptan study group prior to 72 hr time point

CONTACTS AND LOCATIONS:
Overall Officials: Barry E Bleske, Pharm. D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States